CLINICAL TRIAL: NCT04912206
Title: Impact of Emergency Physician-Performed Ultrasound for the Evaluation of Patients With Acute Abdominal Pain, Prospective Randomized Dual Centre Study
Brief Title: Impact of Emergency Physician-Performed Ultrasound for the Evaluation of Patients With Acute Abdominal Pain
Acronym: EchoPAIN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Departemental Vendee (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CHD20_0133
Record Dates: First submitted 2021-05-28; First posted 2021-06-03 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Abdominal Pain
Keywords: Abdominal Pain; Point-of-Care Ultrasound
MeSH Terms: conditions — Abdominal Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Point-of-Care Ultrasound on top of diagnosis work-up
  Interventions: Diagnostic Test: Point-of-Care Ultrasound
- Control (No Intervention): Usual diagnosis work-up without Point-of-Care Ultrasound

INTERVENTIONS:
Diagnostic Test: Point-of-Care Ultrasound — Abdominal clinician-performed Ultrasound
  Arms: Intervention

SUMMARY:
Non-traumatic abdominal pain is one of the most frequent complaints in Emergency Medicine. Point-of-Care Ultrasound (POCUS) has good performance in these situations. It is performed at the patient's bedside with immediate results. It has been demonstrated that a clinician-performed ultrasound was able to increase the diagnosis accuracy in patients with acute abdominal pain. However, the level of evidence of its diagnostic efficacy remains controversial in particular in Europe.

The principal investigators thus aimed to investigate the efficacy of early POCUS on diagnostic accuracy in the context of of non-traumatic abdominal pain by a randomized control study conducted in two emergency departments (ED). Secondary objectives will be comparison between the two groups for time spent in the ED before diagnosis and disposition (discharged home or hospitalization), prescription of complementary examinations and in particular, radiologic exams.

DETAILED DESCRIPTION:
Non-traumatic abdominal pain is one of the most frequent complaints in Emergency Medicine. Point-of-Care Ultrasound (POCUS) has good performance in these situations. It is performed at the patient's bedside with immediate results. It has been demonstrated that a clinician-performed ultrasound was able to increase the diagnosis accuracy in patients with acute abdominal pain.

The principal investigators thus aimed to investigate the efficacy of early POCUS on diagnostic accuracy in the context of of non-traumatic abdominal pain by a randomized control study conducted in two ED. Secondary objectives will be comparison between the two groups for time spent in the ED before diagnosis and disposition (discharged home or hospitalization), prescription of complementary examinations and in particular, radiologic exams.

It will be a randomized, controlled, open and interventional study. In the control group, the diagnosis will be established after clinical examination and reception of biological analysis results. In the interventional group, a POCUS performed in the ED by a local investigator will be added and the diagnosis will be established after clinical exam, biological analysis reception and POCUS. POCUS will only be performed by physicians who have completed a validated training program.

Furthermore, before study initiation, refresh sessions focused on acquisition techniques and pathological findings will be organized in the two participating ED. Such refresher courses were efficient to increase the overall confidence of operators

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years
* Admitted for acute abdominal pain lasting for less than 5 days
* Availability in the ED at that time of an Emergency Physician trained in POCUS
* Patient able to understand the protocol and having given oral informed consent to participate in the study or included under the emergency inclusion procedure

Exclusion Criteria:

* Documented end-of-life with a do-not-resuscitate order
* Immediate need for management for hemodynamic stabilization
* Patient sent to the ED by an out-of-hospital practitioner
* Pregnant and breast-feeding women
* No social security
* Under guardianship, curatorship or deprived of liberty.
* Do not understand French

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 256 (Actual)
Dates: Start 2021-06-11 (Actual); Primary Completion 2022-06-23 (Actual); Study Completion 2022-06-23 (Actual)

PRIMARY OUTCOMES:
Exact diagnostic rate | The reference diagnosis will be determined by an adjudication committee on the basis of an exhaustive analysis of the patient's file at Day 28
  Comparison of the rate of exact diagnostic after clinical exam and biological results with point-of-care ultrasound (interventional arm) or without (control arm) according to the adjudication committee diagnostic (reference diagnosis).

CONTACTS AND LOCATIONS:
Overall Officials: François Brau, Principal Investigator — CHD Vendée; Philippe Leconte, Principal Investigator — Nantes University Hospital
Locations (2):
- France (2):
  - Centre Hospitalier Departemental Vendée, La Roche-sur-Yon
  - Centre Hospitalier Universitaire de Nantes, Nantes

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Brau F, Papin M, Batard E, Abet E, Frampas E, Le Thuaut A, Montassier E, Le Bastard Q, Le Conte P. Impact of emergency physician performed ultrasound in the evaluation of adult patients with acute abdominal pain: a prospective randomized bicentric trial. Scand J Trauma Resusc Emerg Med. 2024 Feb 26;32(1):15. doi: 10.1186/s13049-024-01182-5. PMID 38409086
- [Derived] Brau F, Martin S, Le Bastard Q, Ricaud P, Legrand A, Montassier E, Le Conte P. Impact of emergency physician-performed ultrasound for the evaluation of patients with acute abdominal pain, prospective randomized dual Centre study: study protocol for a diagnostic trial. Trials. 2022 Sep 24;23(1):804. doi: 10.1186/s13063-022-06755-2. PMID 36153600